CLINICAL TRIAL: NCT00748735
Title: Optimal Definition of Left Ventricular Lead Position in Cardiac Resynchronization Therapy by Myocardial Deformation Imaging
Brief Title: Left Ventricular Lead Position in Cardiac Resynchronization Therapy
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Other Study IDs: MB-2008-CRT
Record Dates: First submitted 2008-09-07; First posted 2008-09-09 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-01

CONDITIONS: Heart Failure
Keywords: cardiac resynchronization therapy; echocardiography; heart failure; left ventricular function; pacing; myocardial deformation imaging; Optimal Definition of Left Ventricular Lead Position in Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A1: heart failure patients undergoing CRT implantation
  Interventions: Procedure: Implantation of a cardiac resynchronization therapy device; Procedure: Echocardiography (myocardial deformation imaging)

INTERVENTIONS:
Procedure: Implantation of a cardiac resynchronization therapy device
Procedure: Echocardiography (myocardial deformation imaging)

SUMMARY:
Left ventricular (LV) lead position has crucial impact on cardiac resynchronization therapy (CRT) success. This study will compare fluoroscopy and myocardial deformation imaging for optimal definition of LV lead position.

DETAILED DESCRIPTION:
In a 16 segment model circumferential strain will be used to determine the segment with latest peak systolic circumferential strain prior to CRT, considered as the optimal LV lead target. LV lead will be defined by (1) fluoroscopy, (2) the maximal temporal difference of peak circumferential strain before-to-on CRT and (3) the earliest peak systolic circumferential strain during LV pacing. For all 3 modalities optimal LV lead position is defined as concordance or immediate neighbouring of the segment with defined LV lead position to the determined optimal target segment. At follow-up echocardiography will be performed to determine improvement in LV function and remodeling.

ELIGIBILITY:
Inclusion Criteria:

* See above
* Males and females
* Ages 18 to 80 years

Exclusion Criteria:

* Patients who already have had a pacemaker device
* Patients with poor echocardiographic window
* Patients who are not able to understand the study and to give informed written consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with end-stage heart failure and sinus rhythm, scheduled for new implantation of a biventricular pacemaker were included in the study. Criteria for CRT implantation were New York Heart Association (NYHA) functional class III (N=35) or IV (N=21) despite optimal pharmacologic therapy and evidence of LV systolic dysfunction with ejection fraction <35% and a QRS >120ms.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)

PRIMARY OUTCOMES:
Improvement in LV function and LV remodelling | 6 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Becker, MD, Principal Investigator — RWTH Aachen University Hospital; Rainer Hoffmann, MD, Study Chair — RWTH Aachen University Hospital
Locations (1):
- Department of Cardiology, RWTH Aachen University Hospital, Aachen, Germany

REFERENCES:
- [Background] Becker M, Franke A, Breithardt OA, Ocklenburg C, Kaminski T, Kramann R, Knackstedt C, Stellbrink C, Hanrath P, Schauerte P, Hoffmann R. Impact of left ventricular lead position on the efficacy of cardiac resynchronisation therapy: a two-dimensional strain echocardiography study. Heart. 2007 Oct;93(10):1197-203. doi: 10.1136/hrt.2006.095612. Epub 2007 Feb 19. PMID 17309913
- [Background] Becker M, Kramann R, Franke A, Breithardt OA, Heussen N, Knackstedt C, Stellbrink C, Schauerte P, Kelm M, Hoffmann R. Impact of left ventricular lead position in cardiac resynchronization therapy on left ventricular remodelling. A circumferential strain analysis based on 2D echocardiography. Eur Heart J. 2007 May;28(10):1211-20. doi: 10.1093/eurheartj/ehm034. Epub 2007 Apr 10. PMID 17426079
- [Derived] Becker M, Altiok E, Ocklenburg C, Krings R, Adams D, Lysansky M, Vogel B, Schauerte P, Knackstedt C, Hoffmann R. Analysis of LV lead position in cardiac resynchronization therapy using different imaging modalities. JACC Cardiovasc Imaging. 2010 May;3(5):472-81. doi: 10.1016/j.jcmg.2009.11.016. PMID 20466342